CLINICAL TRIAL: NCT06657313
Title: Is Vitamin D Deficiency Linked to Functional Constipation In Children
Status: Active, not recruiting | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Amany Mohammed El-Rebigi, MD, Amany Mohammed El-Rebigi, Benha University
Other Study IDs: Rc 18-5-2024
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Functional Constipation in Children
Keywords: Vitamin D Deficiency; Functional constipation; Children
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Serum 25-hydroxy vitamin D levels will be measured in patients and healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Constipation is one of the most common causes of patient visits to pediatric clinics. Prevalence of constipation is estimated between 1.9-27.2% in the USA (Rasquin et al., 2006).

In children aged <18 years, its prevalence was about 0.7-29.6%. Untreated constipation may cause fecal impaction and fecal soiling5 which are seen in about 1-3% of children (Bulloch and Tenenbein, 2002).

Constipation may cause gastrointestinal problems such as abdominal pain, anal pruritus, rectal bleeding, and anorexia or non-gastrointestinal complications such as urinary problems (Dehghani et al., 2015).

Functional constipation is defined as constipation without an organic etiology and is diagnosed according to the Rome criteria1-3. The symptom- based Rome criteria were first developed for adults in 1989 during a consensus meeting of experts in the field of functional gastrointestinal disorders. These criteria have been updated several times and are now internationally acknowledged and used for both research and clinical purposes. The revised Rome IV criteria- for childhood and adult functional constipation were published in 2016 (Benninga et al., 2016), (Hyams et al., 2016), (Lacy et al., 2016).

Functional constipation, a common disorder in all age groups, shows some similarities in children and adults, but important differences exist regarding epidemiology, symptomatology, pathophysiology, diagnostic workup and therapeutic management. In this research, we hypothesized that serum vitamin D deficiency could be associated with chronic functional constipation in children secondary to delayed transit intestinal time and consequently we will investigate this relationship and the related psychological aspects.

DETAILED DESCRIPTION:
In this research, we hypothesized that serum vitamin D deficiency could be associated with chronic functional constipation in children secondary to delayed transit intestinal time and consequently we will investigate this relationship and the related psychological aspects.

ELIGIBILITY:
Inclusion Criteria:

- All pediatric Patients from 6 to 16 years old who were diagnosed with chronic constipation in gastrointestinal and hepatology clinic, at Benha university Hospital according to revised Rome IV criteria will be consecutively recruited in this study.

Sex- and age-matched approximate-health children will be recruited as a control group.

Exclusion Criteria:

* 1)- Age < 6 years and > 16 years old. 2)- Children with any chronic medical disease. 3)- Children who receive any medications. 4)- Children with organic causes of constipation such as anal fissure, stenosis or stricture, inflammatory bowel disease and intestinal malabsorption.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All pediatric patients who were diagnosed with chronic functional constipation according to Revised Rome IV criteria included in this study will be subjected to:
  * Demographic data upon admission including age, sex, weight, length, BMI, level of education of parents & residency.
  * The following data will be collected from patients with chronic constipation: Nutritional history, frequency of defecation per day, history of painful or hard bowel movements, history of excessive stool retention, history of large diameter stools, presence of a large fecal mass in the rectum, history of fecal incontinence per week, history of large diameter stools that can obstruct the toilet, duration of the disease and treatment.
  * Clinical data including symptoms as constipation, abdominal pain and swelling and signs like abdominal distension.
  Diagnosis of Functional chronic constipation in pediatric was done according to the Revised Rome IV criteria
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Vitamin D level in Children with functional constipation | 6 months
  Investigate the relationship between serum 25-hydroxyvitamin D levels and functional chronic constipation in children.

CONTACTS AND LOCATIONS:
Overall Officials: Amany M. El-Rebigi, PhD, MD, Principal Investigator — lecturer of pediatric and neonatology, Faculty of medicine, Benha University; Rasha M. Zakaria, PhD, MD, Principal Investigator — lecturer of pediatric and neonatology, Faculty of medicine, Benha University
Locations (1):
- Benha University, Banhā, Al-Qalyubia, Egypt

IPD SHARING:
Plan to Share IPD: No